CLINICAL TRIAL: NCT05123911
Title: A Single Center, Open Label, Safety in Use Clinical Study to Assess the Topical Tolerability and Influence of Routine Use of 3 Investigational Products on the Microbiome and Scalp Attributes in Children With Curly Hair
Brief Title: A Study of 3 Investigational Products on the Microbiome and Scalp Attributes in Children With Curly Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCSSKB004136; CCSSKB004136 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-11-09; First posted 2021-11-17 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Product Kit: Shampoo, Conditioner and Combining Cream (Investigational Products [IPs]) (Experimental): The parents/legally acceptable representative (LAR) of the participants will receive a product kit containing the 3 investigational products (shampoo, conditioner and combining cream) and will bathe the child participant with shampoo followed by conditioner and then apply combining cream to wet and previously moistened hair at least 3 times a week for up to 28 days.
  Interventions: Other: Investigational Shampoo; Other: Investigational Conditioner; Other: Investigational Combing Cream

INTERVENTIONS:
Other: Investigational Shampoo — Parent/LAR will bathe the child participant with the investigational shampoo at least 3 times a week for up to 28 days.
Other: Investigational Conditioner — Parent/LAR will bathe the child participant with the investigational conditioner at least 3 times a week for up to 28 days.
Other: Investigational Combing Cream — Parent/LAR will apply investigational combining cream to wet and previously moistened hair at least 3 times a week for up to 28 days.

SUMMARY:
The purpose of this study is to evaluate the topical safety (tolerability/acceptability) of a kit of cosmetic products (shampoo, conditioner, and combing cream), the presence of residues on the scalp through visual assessment and image capture, the skin barrier, pH, and sebum level. All these evaluations will be performed before and after 28 plus minus (+-) 2 days of use under normal conditions, under the supervision of dermatologist and pediatrician.

ELIGIBILITY:
Inclusion Criteria:

For children

* Female and male children participants
* 3 to 6 years old
* Fitzpatrick Skin Type IV to VI
* Generally, in good health based on medical history reported by the parent/legally acceptable representative (LAR)
* Intact skin in the test region, scalp, (except for the presence of mild seborrheic dermatitis, if applicable)
* Children participants with curly to kinky hair
* Children participants with a minimum hair length of 5 cm (3 fingers)
* Minors under the age of assent should be accompanied by a LAR who can read, write, speak, and understand Portuguese

For parent/LAR of participants

* 18 to 65 years old
* Generally, in good health based on medical history
* Has presented proof of guardianship for the infant participant (that is, birth certificate along with valid Identity document [ID] of parents/LAR)
* Able to read, write, speak, and understand Portuguese
* Individual has signed the informed consent document (ICD) and ICID (Informed consent image document)
* Be willing and able to participate and comply with the study that requires the use of the principal investigator (PIs) as indicated on the child throughout the study period
* Agrees not to use the provided products on any other family member (other than the child participant) for the duration of the study
* Agrees to bathe your child in the shower instead of the bathtub
* Intends to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

For Children

* Has known allergies or adverse reactions to common topical skincare products, including shampoo, conditioner and combing cream
* Presents with a skin condition that may confound the study results (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema or active skin cancer)
* Presents with primary/secondary lesions (example: scars, ulcers, vesicles) on test sites
* Has parent/LAR reported Type 1 or Type 2 diabetes in the participant or is taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including: a) Immunosuppressive or steroidal drugs within 2 months before Visit 1; b) Non-steroidal anti-inflammatory drugs within 5 days before Visit 1; c) Antihistamines within 2 weeks before Visit 1; d) Topical or systemic antibiotics or antifungals within 30 days before Visit 1
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Having had chemical treatments that transform the hair shaft (for example: straightening, hair relaxation, Et cetera [etc.])
* Present folliculitis and/or hair loss disorders
* Use anti-hair loss treatment for at least three months before the study start
* Use anti-dandruff shampoos on the scalp and/or hair for at least three weeks before the study start
* Be using or have used in the last 4 weeks long hairstyles, such as Nago braids made only on natural hair or with the addition of synthetic fiber threads (example: Kanekalon, Jumbo or wool)
* Exposure or having been exposed in the last 7 days to the beach, swimming pool and intense sun during the study period
* Simultaneously participating in any other clinical study
* Be an immediate family member of the PI, Study Site, or Sponsor
* Initiate probiotic treatment or supplementation (Culturelle, Provance, Colidis, Probioatop, Bifidobacterium, Lactobacillus, etc.) during the study
* Change treatment with probiotics (Culturelle, Provance, Colidis, Probioatop, Bifidobacterium, Lactobacillus, etc.) if the participating child is already using them before the study begins

For parent/LAR of participants

* Has known allergies or adverse reactions to common topical skincare products, including shampoo, conditioner and combing cream
* Has reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including: a) Immunosuppressive or steroidal drugs within 2 months before Visit 1; b) Non-steroidal anti-inflammatory drugs within 5 days before Visit 1; c) Antihistamines within 2 weeks before Visit 1
* Is self-reported to be pregnant or planning to become pregnant during the study
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Is simultaneously participating in any other clinical study
* Is an employee/contractor or immediate family member of the PI, study site, or sponsor

Additional exclusion criteria during Coronavirus Disease 2019 (COVID-19) pandemic

* History of a confirmed COVID-19 infection in the last 30 days
* Contact with COVID-19-infected person within 14 days prior to enrollment
* Any international travel within 14 days prior to enrollment including members in the same household
* Participants with self-reported symptoms within the past 2 weeks: a) Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomachaches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, fever, or chest pain/tightness; b) Temperature greater than or equal to (>=) 38 degree Celsius (°C)/100 degree Fahrenheit (°F), measured; c) Use of fever reducers within 2 days prior to each on-site visit

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 28 +- 2 days in Score of Topical Tolerability of the Participant's Scalp | Baseline (Day 1) to 28 +- 2 days
  Change from baseline to 28 +- 2 days in score of topical tolerability of the participant's scalp will be reported. Topical tolerability of investigational products (shampoo, conditioner and combining cream) will be assessed by clinical assessment of the initial condition of the participant's scalp assessed by the dermatologist based on attributes such as: itching, stinging, burning, irritation, dryness, desquamation, and erythema. The attributes will be evaluated using a 5-point scale (0=none, 1=very mild, 2=mild, 3=moderate, 4=intense).
Change from Baseline to 28 +- 2 days in Score of Scalp Residue Through use of Affected Area Criteria | Baseline (Day 1) to 28 +- 2 days
  Change from baseline to 28 +- 2 days in score of scalp residues through use of affected area criteria will be reported. Scalp residue assessment will be performed by a trained technician using the scalp dandruff counting methodology, using a pre-defined seborrheic dermatitis severity scale, in which the amount of residue will be calculated for the four quadrants of the scalp, through the rating scale for the area affected by the residue (where score of 0=less than 10 percent [%] affected area; 1=10-30% affected area; 2=30-50% affected area; 3=50-70% affected area and 4= more than 70% affected area).
Change from Baseline to 28 +- 2 days in Score of Scalp Residue Through use of Severity Criteria | Baseline (Day 1) to 28 +- 2 days
  Change from baseline to 28 +- 2 days in score of scalp residues will be reported. Scalp residue assessment will be performed by a trained technician using the scalp dandruff counting methodology, using a pre-defined seborrheic dermatitis severity scale, in which the amount of residue will be calculated for the four quadrants of the scalp, through the rating scale for residual severity (where score of 1=small flakes reminding of a white powder; 2=intermediate; 3=large flakes adhering to the scalp, appearing as an irregular surface; 4=intermediate; 5=apparently frozen flakes in the form of yellowish plaques attached to the scalp, some with evidence of exudation or erythema).
Change from baseline to 28 +- 2 days in Scalp Skin Barrier Evaluation | Baseline (Day 1) to 28 +- 2 days
  Scalp skin barrier assessment will be performed by a trained technician through instrumental measurements with the Tewameter TM Nano equipment (Courage-Khazaka Electronic GmbH). The Tewameter TM probe measures the rate of water evaporation from the skin's surface. A decrease in transepidermal water loss (TEWL) values indicates an improvement in the scalp skin barrier.
Change from Baseline to 28 +- 2 days in Scalp Sebumetry Evaluation | Baseline (Day 1) to 28 +- 2 days
  The evaluation of scalp sebumetry will be performed by a trained technician through instrumental measurements with the Sebumeter SM 815 (Courage + Khazaka Electronic GmbH) equipment. The equipment principle is based on the change of a translucent membrane that becomes progressively more transparent as it absorbs substances of a lipidic nature.
Change from Baseline to 28 +-2 days in Scalp Skin pH Evaluation | Baseline (Day 1) to Day 28 +-2 days
  Scalp pHmetry evaluation will be performed by a trained technician through instrumental measurements with the Mettler Toledo S8 Seven 2 Go Portable pH equipment. As the skin, with its excretions, is almost an aqueous solution, the pH measurement evaluates an important characteristic of any aqueous solution: acidity or alkalinity. The pH value lies on a point on the scale from 0 (strongly acidic) to 14 (strongly alkaline), with the value 7 representing neutrality.
Change from Baseline to 28 +- 2 days in Scalp Image Capture | Baseline (Day 1) to Day 28 +- 2 days
  The scalp image will be captured by a trained technician, through the Fotofinder equipment, for registering the possible residues found on the scalp and evaluated by a trained technician.

SECONDARY OUTCOMES:
Change from Baseline to 28 +- 2 days in Scalp Microbiome | Baseline (Day 1) and Day 28 +- 2 days
  The scalp microbiome is composed of a group of microorganisms, including bacteria and fungi, that play an important role on the scalp. To evaluate the type and number of bacteria and fungi present on the surface of the scalp, a sample will be collected on this area using a swab. We will analyze the type and number of microorganisms before and after the investigational products (IPs) regimen. This evaluation will be done through metagenomics, a technique that allow the determination of the different types and quantity of microorganisms present in a specific area. The microbiota reads generated from each participating individual are compared against existing public databases to classify the species present and the number of times each appears in the individual's microbiome in the collected area.
Scalp Microbiome Collection and Metagenomic Analysis | Baseline (Day 1)
  The scalp microbiome is composed of a group of microorganisms, including bacteria and fungi, that play an important role on the scalp. To evaluate the type and number of bacteria and fungi present on the surface of the scalp, a sample will be collected on this area using a swab. We will analyze the type and number of microorganisms before and after the IPs regimen. This evaluation will be done though metagenomics, a technique that allows the determination of the different types and quantity of microorganisms present in a specific area. The microbiota reads generated from each participating individual are compared against existing public databases to classify the species present and the number of times each appears in the individual's microbiome in the collected area.
Change from Baseline to 28 +- 2 days in Quality-of-life Questionnaire | Baseline (Day 1) and Day 28 +- 2 days
  Parents/legally acceptable representative (LAR) of children participants will complete a questionnaire consist of 5 questions to report on the quality of life, health, and other areas of the child's life.
Change from Baseline to 28 +- 2 days in Scalp Hydration Evaluation | Baseline (Day 1) and Day 28 +- 2 days
  The scalp hydration evaluation will be performed by a trained technician through instrumental measurements with the DermaLab USB Moisture Module equipment (Cortex Technology). The equipment is based on conductance principle. The higher the conductance, more amount of water, an increase in free electrons happens, therefore, the higher the hydration of the skin. An increase in conductance values indicates an improvement in hydration.

CONTACTS AND LOCATIONS:
Overall Officials: Mariane M Mosca, Bsc, Principal Investigator — Allergisa Pesquisa Dermato-Cosmética Ltda
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética LTDA, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Agência Nacional De Vigilância Sanitária. Guia para Avaliação de Segurança de Produtos Cosméticos. 2a ed., 2012. Available on <http://www.anvisa.gov.br/cosmeticos/guia/guia_cosmeticos_final_2.pdf> Accessed by: 05 Jan 2017
- [Background] ASSOCIAÇÃO MÉDICA MUNDIAL. Declaração de Helsinque. Princípios Éticos para Pesquisa Médica Envolvendo Participantes Humanos. Available on: <http://www.wma.net/en/30publications/10policies/b3/17c.pdf>. Accessed by: 05 Jan 2017.
- [Background] BRASIL. Ministério da Saúde. RDC nº 466, de 12 de dezembro 2012. Aprova diretrizes e normas regulamentadoras de pesquisas envolvendo seres humanos. Available on: <http://conselho.saude.gov.br/resolucoes/2012/Reso466.pdf>. Accessed by: 05 Jan 2017.
- [Background] Cortex Technology. DermaLab® Combo - technical specifications. Available on: https://cortex.dk/multi-parameter-dermalab-combo/.
- [Background] Courage + Khazaka electronic GmbH. Skin-pH-Meter PH 905: The Measuring Principle. Available on: <http://www.courage-khazaka.de/index.php/en/artikel-work/59-products/scientific/132-skinphmeter.
- [Background] Courage + Khazaka electronic GmbH. Sebumeter® SM 815. The Measuring Principle. Available on: https://courage-khazaka.de/en/scientific-products/efficacy-tests/16-wissenschaftliche-produkte/alle-produkte/151-sebumeter-e.
- [Background] Courage + Khazaka electronic GmbH. Tewameter® TM Nano. The Measuring Principle. Available on: https://courage-khazaka.de/en/scientific-products/efficacy-tests/16-wissenschaftliche-produkte/alle-produkte/157-tewameter-nano-e.
- [Background] De la Mettrie R, Saint-Leger D, Loussouarn G, Garcel A, Porter C, Langaney A. Shape variability and classification of human hair: a worldwide approach. Hum Biol. 2007 Jun;79(3):265-81. doi: 10.1353/hub.2007.0045. PMID 18078200
- [Background] International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use.. ICH harmonized tripartite guideline: Guideline for Good Clinical Practice. J Postgrad Med. 2001 Jan-Mar;47(1):45-50. No abstract available. PMID 11590294
- [Background] OPAS. Organização Pan-Americana de Saúde. Boas Práticas Clínicas: Documento das Américas. IV Conferência Pan-Americana para Harmonização da Regulamentação Farmacêutica, 2005. Disponível em: http://www.anvisa.gov.br/medicamentos/pesquisa/boaspraticas_americas.pdf Acesso em: 10 18 MAR ABR 2016.
- [Background] Saxena R, Mittal P, Clavaud C, Dhakan DB, Roy N, Breton L, Misra N, Sharma VK. Longitudinal study of the scalp microbiome suggests coconut oil to enrich healthy scalp commensals. Sci Rep. 2021 Mar 31;11(1):7220. doi: 10.1038/s41598-021-86454-1. PMID 33790324
- [Background] Oliveira, A. C. S. TRANÇANDO CABELO, IDENTIDADE, ESTIGMA E CONSUMO: um estudo sobre as maneiras de consumir relacionadas à manipulação capilar de mulheres de cabelos crespos e cacheados a partir da teoria da prática. Dissertação (mestrado) - Universidade Federal de Minas Gerais, Centro de Pós-Graduação e Pesquisas em Administração (2019). Disponível em: https://repositorio.ufmg.br/bitstream/1843/30441/1/Disserta%C3%A7%C3%A3o_finalizada%20-%20Ana%20Carolina%20Soares.pdf. Acesso em: 17 SET 2021.
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSSKB004136&attachmentIdentifier=d49ad554-89b1-453f-9cc0-2cc28d828ec6&fileName=Summary_CSR_for_ClinTrials.gov_0130.pdf&versionIdentifier=